CLINICAL TRIAL: NCT05800236
Title: Characterisation of the Intratumoral Microbiome in Gastric Adenocarcinoma: to a Personalised Medicine
Acronym: MICROGAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2022/09
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Gastric Adenocarcinoma
Keywords: Gastric cancer; intratumoral microbiota; circulating tumour cells; biomarkers
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastric adenocarcinoma (Other): patients who undergo gastrectomy
  Interventions: Procedure: Gastrectomy

INTERVENTIONS:
Procedure: Gastrectomy — Patients operated on for curative purposes at the Bordeaux University Hospital for gastric adenocarcinoma of any type or stage and Collection of two venous blood tubes

SUMMARY:
In this study, gastric tumours and adjacent healthy mucosa will be collected from gastric cancer patients operated on for curative purposes. From this material, presence and characterisation of intratumoral bacteria will be determined. Intratumoral microbiota composition will be compared with healthy adjacent tissue, and the intratumoral microbiota composition will also be compared between different tumor types. The different bacterial signatures that we will characterise may be used as biomarkers.

DETAILED DESCRIPTION:
Gastric adenocarcinoma is mainly linked to Helicobacter pylori infection, and this bacterium is classified as a class 1 carcinogen by the WHO. However, infection with this bacterium alone is not sufficient for the development of gastric adenocarcinoma. It is now recognised that environmental factors such as the digestive microbiota influence carcinogenesis. Improved sequencing techniques have shown that some tumours contain intracellular bacteria and that these are specific to the origin of the tumour. A study describing the existence of intratumoral bacteria was carried out on 7 different tumour types excluding gastric cancer. Gastric adenocarcinoma is a cancer with a poor prognosis, treatment, based mainly on surgery combined with conventional chemotherapy, is not very effective with a 5-year survival rate of less than 20%. Except for Her2+ cases, there is no specific treatment. It is therefore now essential to develop targeted and effective treatments.

The objective of this project is to define whether intratumoral bacteria exist in gastric cancer.

To achieve this, tumours and adjacent healthy mucosa from patients with gastric cancer will be collected and analysed in INSERM U1312 laboratory. The biological material studying consists only of remnants of biopsies of gastric tumours and adjacent healthy tissues, which are not needed in the pathology laboratory, from patients who undergo gastrectomy as part of their cancer management Two blood tubes for the isolation of possible circulating tumour cells will also be collected. From these materials, the presence of intratumoral bacteria will be determined by immunohistochemistry targeting components of the bacterial wall, by RNAscope® targeting 16S ribosomal RNA (16S rRNA) and by real-time quantitative PCR targeting 16S rDNA. Characterisation of the intratumoral microbiota will be performed by sequencing 16S rDNA gene. The collected blood will be tested for the presence of CSCs and, if CSCs are detected, the microbiota will be tested and characterised using the same techniques described above.

The primary endpoint will be the evidence of an intratumoral microbiota and its taxonomic description.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated on for curative purposes at the Bordeaux University Hospital for gastric adenocarcinoma of any type or stage
* Histological evidence of gastric adenocarcinoma by biopsies taken at diagnosis
* No oral opposition to participate after being informed about the study
* Beneficiary of a social security scheme
* Major

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient placed under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-22 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Observation of type of intratumoral microbiota by microscopy | Day 1
  Description of intratumoral microbiota in gastric adenocarcinoma, no statistical tests will be necessary.

SECONDARY OUTCOMES:
Detection of bacteria in CTCs | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Emilie BESSEDE, PharmD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Hôpital du Haut Lévêque, Pessac, France